CLINICAL TRIAL: NCT02723721
Title: Prospective Study of Ingenol Mebutate for Non-invasive Lentigo Melanoma of the Face - Study PICAMEL
Brief Title: Prospective Study of Ingenol Mebutate for Non-invasive Lentigo Melanoma of the Face
Acronym: PICAMEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-PP-14
Record Dates: First submitted 2016-03-15; First posted 2016-03-30 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2020-11

CONDITIONS: Lentigo Maligna
Keywords: Lentigo maligna
MeSH Terms: conditions — Hutchinson's Melanotic Freckle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Picato gel (Experimental): application on1 cm around the lesion, 0.47 g of Picato® gel 150 µg/g, once a day on 3 consecutive days.
  Interventions: Drug: Picato gel

INTERVENTIONS:
Drug: Picato gel — apply on and 1 cm around the lesion, 0.47 g of Picato® gel 150 µg/g, once a day on 3 consecutive days.

SUMMARY:
Non-invasive lentigo maligna (LM) is characterized by an in situ proliferation of melanoma cells, limited to the epidermis. It is found most commonly on the head and neck of elderly persons, with a peak incidence in the seventh or eighth decade. If untreated, it may develop into invasive melanoma. The gold standard treatment for LM is surgery using a 5-10 mm margin. However, the lesions can be large, and conventional surgery can be difficult, particularly on the face.

Then, there is a need for a topical non-surgical treatment of LM. Ingenol mebutate (IM)/Picato® is able to induce cell apoptosis and an inflammatory reaction in the epidermis and superficial dermis.

Thus, the investigators hypothesize that the topical use of Picato® could induce the cure or a prolonged remission of non-invasive LM.

Because of the exploratory phase of this study (no case report and no clinical trial at the early phase of designing this study, only one case report at the time of submission of this form) the investigators will conduct an open label study limited to patients who are not eligible to, or who refuse surgical treatment of their LM.

The main objective of this study is to determine the proportion of patients with complete response (CR) obtained 2 months after one or two cycles (for patients who did not respond to the first cycle) of topical treatment by IM 150 µg/g for non-invasive LM of the face (head and neck).

DETAILED DESCRIPTION:
Lentigo maligna (LM) is a form of malignant melanoma in situ seen predominantly on chronically sun-damaged skin. It is found most commonly on the head and neck of elderly persons, with a peak incidence in the seventh or eighth decade. If untreated, it may develop into invasive melanoma. The gold standard treatment for LM is surgery using a 5-10 mm margin. However, the lesions can be large, and conventional surgery can be difficult, particularly on the face. Furthermore, the extent of LM tends to be underestimated because the exact limits of the lesion are not always easy to determine. Thus, relapses and repeated surgical procedures are common. Moreover, LM appears in elderly people who often have anaesthetic contraindications. When surgery is not or no more feasible, superficial radiotherapy or destructive treatment by topical immunotherapy using imiquimod 5% cream may be used, but the efficacy of these treatments remains to be clearly defined. Regarding the use of imiquimod it has been reported in about 15 isolated cases and in 7 open studies (most of them prospective) for a total of 189 patients. The modalities of use were variable but most of the time once a day, 5 days per week for 3 months. The response rate varied from 53 % to 100%. The major limitations to the use of imiquimod are: 1- a possible lower rate of remission than surgery; 2- the observance of a topical irritating treatment for an extended period.

Thus, there is a need for a topical non-surgical treatment of LM.

Picato® is a topical gel for cutaneous application that contains the active substance ingenol mebutate, which is obtained from the aerial parts of the plant species Euphorbia peplus. by extraction and purification. It is indicated for the cutaneous treatment of non-hyperkeratotic, non-hypertrophic actinic keratosis in adults. The mechanism of action of ingenol mebutate in actinic keratosis is not fully understood. In vivo and in vitro models have shown a dual mechanism of action: 1) induction of local lesion cell death and 2) promotion of an inflammatory response characterised by infiltration of immunocompetent cells.

In addition to this effect on actinic keratoses, a recent study has shown that treatment of superficial basal cell carcinomas with ingenol mebutate gel 500 µg/g under occlusion with an aluminum disk, was efficacious, even when applied only for one day. On the contrary, the same treatment for up to 3 consecutive days showed less clinical benefit in seborrheic keratoses, suggesting a selectivity or penetration variations of ingenol mebutate for cancer cells vs benign cells.

In vitro, it has been shown that ingenol mebutate is able to kill melanoma cells mainly by induction of apoptosis which seems to be secondary to the activation of Protein Kinase C. Based on these data and on previous studies with imiquimod, the investigators suggest that ingenol mebutate might have a clinical effect on melanoma, particularly for superficial intraepidermal lesions of LM. Because these lesions are mostly localised on the face, the concentration of 150 µg/g should be tested first to avoid local skin secondary effects.

The investigators hypothesize that the topical use of Picato® will induce the cure or a prolonged remission of non-invasive LM in patients that are not eligible to or refuse surgery.

The main objective of this study is to determine the proportion of patients with complete response (CR) obtained 2 months after one or two cycles (for patients who did not respond to the first cycle) of topical treatment by IM 150 µg/g for non-invasive LM of the face (head and neck).

The secondary objectives are:

1. To assess the disease-free survival after 1 or 2 cycles of IM 150μg / g. for non-invasive LM,
2. To determine the safety of treatment,
3. To evaluate the diagnostic performance of in vivo reflectance confocal microscopy (RCM) and High Definition Optical Coherence Tomography (HD-OCT) for diagnosis of treatment failure and relapse of LM compared to the standard represented by pathological examination, in monitoring of treatment response and relapse.

The patients will be included after providing informed consent if they have a biopsy-proven non-invasive LM on the head (face or scalp) and if they are not eligible to, or if they refuse surgical treatment.

They will apply on and 1 cm around the lesion, 0.47 g of Picato® gel 150 µg/g, once a day on 3 consecutive days.

The short term efficacy will be evaluated at 2 months, clinically (with Wood's lamp and dermoscopic examination) and histopathologically.

For patients being cured at 2 months, the long term efficacy will be evaluated every 6 months for 36 months, using the same criteria.

For patients having no or only partial remission at 2 months, the treatment will be applied using the same protocol (0.47 g of Picato® gel 150 µg/g, once a day on 3 consecutive days on and 1 cm around the lesion). They will be evaluated 2 months after the retreatment and then every 6 months for 36 months. The safety and local side effects will be evaluated at each visit.

For centers equipped with in vivo reflectance confocal microscopy (RCM) and high-definition optical coherence tomography (HD-OCT), patients will have imaging of the lesion with these techniques before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject of both sexes at least 18 years of age
* Patient with a noninvasive LM of the head (face or scalp) which has been proven by biopsy
* LM with a surface area equal or superior to 1 cm2
* Patient who is not eligible to, or refuse surgical treatment
* LM which has not been treated previously or which has already been treated surgically (one or several time) but which is relapsing or which could not been completely removed
* ECOG (Eastern Cooperative Oncology Group) ≤2
* Patient affiliated to French social security
* Patient able to understand and communicate with the investigator and to comply with the requirements of the study
* Patient must give a written, signed and dated informed consent before any study related activity is performed. Where relevant, a legal representative will also sign the informed study consent according to local laws and regulations

Exclusion Criteria:

Location of the LM:

* on the eyelids or within 1 cm of the eyelids
* within 1 cm of the lips
* within 5 cm of an incompletely healed wound
* elsewhere than on the head

  * LM which is not strictly intraepidermal, which has an invasive component on the biopsy performed at screening visit
  * LM which has had in the past an invasive component, even if it has been surgically treated
  * Melanoma of another histopathologic type than LM
  * LM with a surface area to be treated (including the 1cm surrounding normal skin) > 25 cm2
  * LM whose borders cannot be easily defined
  * Known sensitivity or allergy to any of the ingredients in ingenol mebutate gel
  * Patient treated with topical steroids or others immunosuppressives drugs (local or systemic agents) within 30 days of entry into this trial
  * Patient with active malignancy (other than LM) or a previous malignancy within the past 3 years; except for patient with resected basal cell carcinoma, resected cutaneous squamous cell carcinoma , resected carcinoma in-situ of the cervix, and resected carcinoma in-situ of the breast
  * Past medical history record of infection with human immunodeficiency virus
  * Organ transplant recipient
  * Immunosuppressed subject
  * Women of child-bearing potential, or pregnant or lactating
  * History or evidence of skin conditions other than the trial indication that would interfere with evaluation of the trial medication in the selected treatment area (e.g., eczema, unstable psoriasis, xeroderma pigmentosum).
  * Use of ingenol mebutate and/or imiquimod in and within 5 cm of the selected treatment area within 2 years prior to visit 1
  * Use of cosmetic or therapeutic products and procedures which could interfere with the assessments of the treatment area.
  * Current enrolment or participation in a clinical trial within 30 days of entry into this trial
  * Any medical or psychiatric condition which, in the Investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
the clinical and histological complete response (CR) of non-invasive LM 2 months after the end of a treatment cycle. In case of failure of the first cycle, a second will be realized and the CR will be re-assessed at 4.5 months | at 2 months after end of treatment

SECONDARY OUTCOMES:
disease-free survival | maximum of 36 months
  calculated from the date of the CR and the date of relapse or death related to the non-invasive LM (very unlikely here). Relapse is defined as the clinical appearance of a new pigmented lesion with histopathological analysis, from one or more biopsy (s), which confirms the diagnosis of non-invasive LM.
side effects | at 36 months
  • The type, frequency, severity and the time to onset of side effects will be reported. The side effects will be classified into grades according to WHO criteria and also using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The intensity of short-term local side effects will be evaluated by the Local Skin Reaction score
specific diagnostic signs of treatment failure | maximun of 36 months
relapse of non-invasive LM | maximum of 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Henri MONTAUDIE, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (8):
- France (8):
  - AP-HP Hopital Avicenne, Bobigny
  - AP-HP Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital du Morvan, Brest
  - CHRU de Lille, Lille
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - Hôpital Pontchaillou, Rennes
  - CHU de Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No